CLINICAL TRIAL: NCT02797821
Title: A Phase 2a, Randomized, Multicenter, Open-Label, Pharmacokinetic, and Dose Response Study of Asfotase Alfa in Adult Patients With Pediatric-Onset Hypophosphatasia
Brief Title: Pharmacokinetic and Dose Response Study of Asfotase Alfa in Adult Patients With Pediatric-Onset Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA-HPP-208
Record Dates: First submitted 2016-05-23; First posted 2016-06-14 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Hypophosphatasia
Keywords: HPP; asfotase alfa
MeSH Terms: conditions — Hypophosphatasia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Asfotase Alfa 0.5 mg/kg Dose (Experimental): Participants received 0.5 milligrams (mg) per kilogram (kg) of asfotase alfa administered subcutaneously (SC) 3 times a week from Weeks 3 through 9 following the initial single dose on Day 1 in Week 1.
  Interventions: Drug: Asfotase alfa
- Asfotase Alfa 2.0 mg/kg Dose (Experimental): Participants received 2.0 mg/kg of asfotase alfa administered SC 3 times a week from Weeks 3 through 9 following the initial single dose on Day 1 in Week 1.
  Interventions: Drug: Asfotase alfa
- Asfotase Alfa 3.0 mg/kg Dose (Experimental): Participants received 3.0 mg/kg of asfotase alfa administered SC 3 times a week from Weeks 3 through 9 following the initial single dose on Day 1 in Week 1.
  Interventions: Drug: Asfotase alfa

INTERVENTIONS:
Drug: Asfotase alfa
  Other Names: Strensiq

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of asfotase alfa in adult participants with pediatric-onset HPP.

ELIGIBILITY:
Inclusion Criteria:

1. Participants or their legal representative(s) provided written informed consent prior to undergoing any study-related procedures.
2. Participants were ≥18 years of age at Screening.
3. Participant had pediatric-onset hypophosphatasia (HPP), defined as onset of first sign(s)/symptom (s) of HPP prior to 18 years of age.
4. Participants had a documented diagnosis of HPP as indicated by a documented history of HPP-related skeletal abnormalities and 1 or more of the following:

   * Documented tissue-nonspecific alkaline phosphatase (TNSALP) gene mutation(s) from a certified laboratory.
   * Serum alkaline phosphatase (ALP) level below the age-adjusted normal range AND plasma pyridoxal-5'-phosphate (PLP) above the upper limit of normal at Screening.
5. Participants had a plasma inorganic pyrophosphate (PPi) level of ≥3.9 micromolar (µM) at Screening.
6. Female participants of childbearing potential had a negative pregnancy test at the time of enrollment.
7. Sexually active male and female participants of childbearing potential agreed to use a highly effective method of birth control during the study.
8. Female participants not of child-bearing potential due to sterilization (at least 6 weeks after surgical bilateral oophorectomy with or without hysterectomy or at least 6 weeks after tubal ligation) confirmed by medical history, or menopause.
9. Participants were willing to comply with study procedures and the visit schedule.

Exclusion Criteria:

1. Investigational site personnel directly affiliated with this study and/or their immediate families. Immediate family was defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
2. Employees of Alexion Pharmaceuticals.
3. Currently enrolled in a clinical study involving another study drug or non-approved use of a drug or device.
4. Participated, within the last 30 days, in a clinical study involving a study drug (other than the study drug used in this study).
5. Completed or withdrawn from this study or any other study investigating asfotase alfa in the previous 3 years.
6. Women who were pregnant, planning to become pregnant, or breastfeeding.
7. Serum 25-hydroxy Vitamin D levels below 20 nanogram (ng) per milliliter (mL) at Screening.
8. Screening serum creatinine or parathyroid hormone (PTH) levels ≥1.5 times the upper limit of normal.
9. Any medical condition, serious concurrent illness and/or injury, recent orthopedic surgery, or other extenuating circumstance that, in the opinion of the Investigator, may have significantly interfered with study compliance or study endpoints.
10. Prior treatment with bisphosphonates within 2 years of study entry for any length of time or for more than 2 consecutive years at any prior timepoint.
11. Treatment with PTH, strontium, or sclerostin inhibitors within 6 months prior to the first dose of study drug.
12. Unwilling or unable to comply with the use of a data collection device on which study participants directly recorded data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Shriners Hospitals for Children, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt Medical Center Endocrinology, Nashville, Tennessee
- University of Würzburg, Würzburg, Germany

REFERENCES:
- [Derived] Pan WJ, Pradhan R, Pelto R, Seefried L. Pharmacokinetics of Asfotase Alfa in Adult Patients With Pediatric-Onset Hypophosphatasia. J Clin Pharmacol. 2021 Oct;61(10):1334-1343. doi: 10.1002/jcph.1870. Epub 2021 Jun 19. PMID 33822385
- [Derived] Seefried L, Kishnani PS, Moseley S, Denker AE, Watsky E, Whyte MP, Dahir KM. Pharmacodynamics of asfotase alfa in adults with pediatric-onset hypophosphatasia. Bone. 2021 Jan;142:115664. doi: 10.1016/j.bone.2020.115664. Epub 2020 Sep 26. PMID 32987199
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asfotase Alfa 0.5 mg/kg Dose | Asfotase Alfa 2.0 mg/kg Dose | Asfotase Alfa 3.0 mg/kg Dose
Started | 8 | 10 | 9
Received at Least 1 Dose of Study Drug | 8 | 10 | 9
Completed | 8 | 10 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): randomized participants who received ≥1 dose of study drug and had ≥1 pretreatment and ≥1 on-treatment inorganic pyrophosphate (PPi) result.
Groups:
- Asfotase Alfa 0.5 mg/kg Dose: Participants received 0.5 mg/kg of asfotase alfa administered SC 3 times a week from Weeks 3 through 9 following the initial single dose on Day 1 in Week 1.
- Total: Total of all reporting groups
Arm/Group | Asfotase Alfa 0.5 mg/kg Dose | Asfotase Alfa 2.0 mg/kg Dose | Asfotase Alfa 3.0 mg/kg Dose | Total
Number analyzed (Participants) | 8 | 10 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (17.90) | 42.7 (16.77) | 50 (17.01) | 44.8 (16.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 3 | 4 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 10 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 10 | 9 | 26
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Inorganic Pyrophosphate (PPi) [Mean (Standard Deviation); unit: μM (micromolar)] | 5.4 (1.64) | 5.3 (1.22) | 5 (0.86) | 5.2 (1.23)
Baseline Pyridoxal 5'-Phosphate (PLP) [Mean (Standard Deviation); unit: nanogram (ng)/milliliter (mL)] | 309.5 (349.16) | 382.1 (385.89) | 229.5 (321.43) | 309.7 (346.99)

OUTCOME MEASURES:

1. Primary Outcome: Change In Plasma PPi From Baseline To Pre-3rd Dose At Week 9
Description: Plasma PPi concentrations were determined using a specific enzyme-catalyzed reaction with a radiolabelled marker in a 3-step process. Baseline plasma PPi values were calculated by averaging pre-dose values from samples collected during the Run-in Period at -168, -156, -24, -12, and 0 hours before Baseline. Week 9 plasma PPi values were calculated using blood samples collected before administration of the 3rd dose. The analysis was a restricted maximum likelihood (REML)-based repeated measures mixed model with treatment, visit, sex, Baseline PPi, Baseline weight group (≥ median versus < median), and study drug lot assignment as factors, and an unstructured covariance structure for within-participant correlation.
  Per inclusion criteria, participants had to have had a Screening PPi concentration of ≥3.9 micromolar (μM). Three participants (1 in each group) had Screening PPi concentrations of ≥3.9 μM, but Baseline PPi values ranged between 3.5 to 3.8 μM.
Time Frame: Baseline to Week 9
Population: FAS: randomized participants who received ≥1 dose of study drug and had ≥1 pretreatment and ≥1 on-treatment PPi result.
Measure: Least Squares Mean (Standard Error); unit: μM
Arm/Group | Asfotase Alfa 0.5 mg/kg Dose | Asfotase Alfa 2.0 mg/kg Dose | Asfotase Alfa 3.0 mg/kg Dose
Number analyzed (Participants) | 8 | 10 | 8
μM | -2.604 (0.2399) | -3.797 (0.1949) | -4.484 (0.2120)
Statistical Analysis 1: Comparison: Asfotase Alfa 0.5 mg/kg Dose vs Asfotase Alfa 3.0 mg/kg Dose; A fixed sequence testing procedure was performed to compare the 3.0 mg/kg cohort with the 0.5 mg/kg cohort first. The hypothesis testing for the second comparison of the 2.0 mg/kg cohort compared with the 0.5 mg/kg cohort was only performed if the null hypothesis was rejected for the previous comparison at a significance level of 0.05 (p-value <0.05). The primary endpoint was met if the null hypothesis was rejected for both comparisons at a significance level of 0.05 (both p-values <0.05); Test type: Other; p < 0.0001, REML — REML-based repeated measures mixed model (treatment, visit, sex, Baseline PPi, Baseline weight group [≥median vs < median], and study drug lot assignment as factors) with an unstructured covariance structure for within-participant correlation; A fixed sequence testing procedure was used to control the Type I error rate. A statistical adjustment of p-values was not performed; Least Squares (LS) Means Difference = -1.880, 95% CI 2-sided [-2.544 to -1.216]
Statistical Analysis 2: Comparison: Asfotase Alfa 0.5 mg/kg Dose vs Asfotase Alfa 2.0 mg/kg Dose; A fixed sequence testing procedure was performed to compare the 3.0 mg/kg cohort with the 0.5 mg/kg cohort first. The hypothesis testing for the second comparison of the 2.0 mg/kg cohort compared with the 0.5 mg/kg cohort was only performed if the null hypothesis was rejected for the first comparison at a significance level of 0.05 (p-value <0.05). The primary endpoint was met if the null hypothesis was rejected for both comparisons at a significance level of 0.05 (both p-values <0.05); Test type: Other; p = 0.0008, REML — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Means Difference = -1.193, 95% CI 2-sided [-1.805 to -0.581]

2. Secondary Outcome: Change In Plasma PLP From Baseline To Pre-3rd Dose At Week 9
Description: Plasma PLP was quantified using liquid chromatography/mass spectrometry. Baseline plasma PLP values were calculated by averaging the pre-dose PLP values from blood samples collected during the Run-in Period at -168, -156, -24, -12, and 0 hours before Baseline. Week 9 PLP values were calculated using blood samples collected before the administration of the 3rd dose. The analysis was a REML-based repeated measures mixed model with treatment, visit, sex, Baseline PPi, Baseline weight group (≥ median versus < median) and study drug lot assignment as factors, and an unstructured covariance structure for within-participant correlation.
Time Frame: Baseline to Week 9
Population: FAS: randomized participants who received ≥1 dose of study drug and had ≥1 pretreatment and ≥1 on-treatment PPi result.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Asfotase Alfa 0.5 mg/kg Dose | Asfotase Alfa 2.0 mg/kg Dose | Asfotase Alfa 3.0 mg/kg Dose
Number analyzed (Participants) | 8 | 10 | 9
ng/mL | -303.955 (9.4075) | -333.447 (8.1486) | -338.002 (85145)
Statistical Analysis 1: Comparison: Asfotase Alfa 0.5 mg/kg Dose vs Asfotase Alfa 3.0 mg/kg Dose; Test type: Other; p = 0.0128, Restricted maximum likelihood-based — REML-based repeated measures mixed model (treatment, visit, sex, Baseline PPi, Baseline weight group [≥ median versus < median], and study drug lot assignment as factors) with an unstructured covariance structure for within-participant correlation; A statistical adjustment of p-values was not performed; LS Means Difference = -34.047, 95% CI 2-sided [-60.171 to -7.922]
Statistical Analysis 2: Comparison: Asfotase Alfa 0.5 mg/kg Dose vs Asfotase Alfa 2.0 mg/kg Dose; Test type: Other; p = 0.0239, Restricted maximum likelihood-based — [p-value comment as in outcome 2, analysis 1]; A statistical adjustment of p-values was not performed; LS Means Difference = -29.492, 95% CI 2-sided [-54.723 to -4.261]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were monitored continuously throughout the study, from the run-in period through the safety follow-up call, which occurred 90 days after the last dose of study drug.
Description: Results for AEs occurred in >5% of the overall Safety population. An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, biologic, or medical device, which did not necessarily have a causal relationship with the asfotase alfa.
Groups:
- Asfotase Alfa 0.5 mg/kg Dose: Participants received 0.5 mg/kg of asfotase alfa administered SC 3 times a week (1 dose each on Mondays, Wednesdays, and Fridays) from Weeks 3 through 9 following the initial single dose on Day 1 in Week 1.
- Asfotase Alfa 2.0 mg/kg Dose: Participants received 2.0 mg/kg of asfotase alfa administered SC 3 times a week (1 dose each on Mondays, Wednesdays, and Fridays) from Weeks 3 through 9 following the initial single dose on Day 1 in Week 1.
- Asfotase Alfa 3.0 mg/kg Dose: Participants received 3.0 mg/kg of asfotase alfa administered SC 3 times a week (1 dose each on Mondays, Wednesdays, and Fridays) from Weeks 3 through 9 following the initial single dose on Day 1 in Week 1.
Arm/Group | Asfotase Alfa 0.5 mg/kg Dose | Asfotase Alfa 2.0 mg/kg Dose | Asfotase Alfa 3.0 mg/kg Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asfotase Alfa 0.5 mg/kg Dose (N=8) | Asfotase Alfa 2.0 mg/kg Dose (N=10) | Asfotase Alfa 3.0 mg/kg Dose (N=9)
Fatigue (General disorders) | 3 | 4 | 3
Injection site erythema (General disorders) | 2 | 3 | 4
Injection site reaction (General disorders) | 1 | 3 | 4
Injection site pain (General disorders) | 2 | 1 | 3
Pain (General disorders) | 1 | 2 | 1
Feeling hot (General disorders) | 0 | 1 | 2
Influenza like illness (General disorders) | 1 | 0 | 1
Injection site bruising (General disorders) | 1 | 0 | 1
Injection site discomfort (General disorders) | 0 | 1 | 1
Injection site haematoma (General disorders) | 2 | 0 | 0
Peripheral swelling (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 3 | 3 | 5
Paraesthesia (Nervous system disorders) | 0 | 0 | 4
Disturbance in attention (Nervous system disorders) | 1 | 0 | 1
Head discomfort (Nervous system disorders) | 1 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 3
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 2
Restlessness (Psychiatric disorders) | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT02797821/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT02797821/SAP_001.pdf